CLINICAL TRIAL: NCT00843232
Title: Physiopathology of Type 2 Diabetes Initiated After Sixty Years Old: Characterization of a Diabetic-related Incretinpathy in Aging Subjects.
Brief Title: Characterization of the Incretinpathy in Type 2 Diabetes Initiated After Sixty Years Old
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Bruno Geloneze, University of Campinas, Brazil
Other Study IDs: LIMED0007
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: diabetes mellitus, type 2; Insulin resistance; Aging; Incretins; DPP-IV protein, human; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; insulin; glucagon; ghrelin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sera and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Elderly T2DM: Elderly T2DM subjects 65 to 80 years old
- Middle-age T2DM: Middle-age T2DM subjects 35 to 50 years old

SUMMARY:
Type 2 diabetes (T2DM) is characterized by hyperglycemia, insulin resistance, absolute or relative insulin deficiency, hyperglucagonemia, increased hepatic glucose production, frequently accelerated gastric emptying and obesity. The known effects of the incretin hormone glucagon-like peptide-1 (GLP-1) on the metabolism are stimulation of insulin secretion, inhibition of glucagon secretion and hepatic glucose production, reduction in gastric emptying and modulation of the appetite. T2DM have disturbances in this system, providing a rationale for therapeutic use of GLP-1 in T2DM. Furthermore, GLP-1 seems to exert trophic effects on the beta-cell.

Dipeptidyl Peptidase IV (DPP-IV) inhibitors represent a new class of oral anti-hyperglycemic agents for the treatment of T2DM. The therapeutic utility of these antihyperglycemic agents rests on their ability of to increase active (intact) levels of incretin peptides, including GLP-1 and GIP.

Twenty four T2DM volunteers will be evaluated by a meal tolerance test (MTT) for incretin hormone measurements, and by the hyperglycemic clamp followed by an arginine test for assessing the beta-cell function and the acute insulin response. Others parameters as body composition and basic biochemistry will be also evaluated at Laboratory of Investigation on Metabolism and Diabetes - LIMED / State university of Campinas, Brazil.

T2DM in elderly are behaving differently. Elderly patients have no increase in liver production of glucose; when obese, have normal insulin secretion, however, display extreme resistance to its action. In non obese individuals, the concentration of glucose necessary for insulin secretion is increased and the action is standard. These findings suggest therefore that the approach should be differentiated treatment for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Stable weight (<5% variation) within the last three months
* Age: 35 to 50 years old for middle-age group, and 65 to 80 y old for elderly group
* Body mass index (BMI): 20 to 29.9kg/m2
* T2DM with diagnosis above 35 years and less than 5 years (Middle-age group)
* T2DM with diagnosis above 65 years and less than 5 years (Elderly group)
* Use of oral antidiabetic drugs (that must at stable dose within the last 3 months)
* Not have participated in any study of intervention with drugs in the last six months.

Exclusion Criteria:

* Use of estrogen, progestogen, active antipsychotics and systemic corticosteroids
* Use of DPP-IV inhibitors and incretin mimetics (current or within 1 month before)
* Continuous use of insulin or glitazone
* Hepatic cirrhosis, renal failure or any clinical condition with impaired insulin sensitivity
* Smoking
* Obesity
* Uncontrolled systemic or disabling diseases
* T2DM treated by non pharmacological methods
* Patients submitted to bariatric surgery
* Latent autoimmune diabetes of the adult (positive anti-GAD antibodies)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Type 2 Diabetes subjects
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Distinctive curves of glucose, C peptide, insulin, glucagon, GLP-1, GIP and ghrelin during a standardized mixed meal tolerance test, in T2DM subjects after sixty-five years old in comparison with middle-age T2DM subjects | within 1 month from screening visit

SECONDARY OUTCOMES:
Distinctive whole-body insulin sensitivity, as estimated by hyperglycemic clamp in T2DM subjects after sixty-five years old in comparison with middle-age T2DM subjects. | within 1 month from screening visit
Distinctive beta-cell function (beta-cell secretion and sensitivity), as measured by hyperglycemic clamp, in T2DM subjects after sixty-five years old in comparison with middle-age T2DM subjects | within 1 month from screening visit
Distinctive acute insulin response as measured by arginine stimulation test in T2DM subjects after sixty-five years old in comparison with middle-age T2DM subjects. | within 1 month from screening visit
Distinctive DPP-IV activity as measured by spectrophotometer in T2DM subjects after sixty-five years old in comparison with middle-age T2DM subjects. | within 1 month from screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Geloneze, MD, PhD, Principal Investigator — LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP); José Carlos Pareja, MD, PhD, Principal Investigator — LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP); Carla Fiori, Nurse, Principal Investigator — LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP); Marcelo MO Lima, MD, Principal Investigator — LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP); Ana Carolina Vasques, MSNutr, Principal Investigator — LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP), Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Geloneze B, de Oliveira Mda S, Vasques AC, Novaes FS, Pareja JC, Tambascia MA. Impaired incretin secretion and pancreatic dysfunction with older age and diabetes. Metabolism. 2014 Jul;63(7):922-9. doi: 10.1016/j.metabol.2014.04.004. Epub 2014 Apr 12. PMID 24854384